CLINICAL TRIAL: NCT01354418
Title: A Randomized Crossover Bioequivalence Study Comparing a Single Dose of Phenylephrine HCl 30 mg Extended Release Tablet to Three Phenylephrine HCl 10 mg Immediate Release Tablets Each Consecutively Dosed Four Hours Apart Under Fed and Fasting Conditions
Brief Title: Bioequivalence of Single Dose Phenylephrine Extended Release Tablets and Phenylephrine HCl Immediate Release Tablets Dosed Every Four Hours (P08340)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18124; CL2010-18 (Other: Protocol Number); P08340 (Other: Merck)
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Nasal Congestion
MeSH Terms: conditions — Nasal Obstruction | interventions — Oxymetazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phenylephrine HCl Extended Release - Fasted (Experimental): Single dose phenylephrine HCl extended release tablet administered under fasted conditions on Day 1 in one of four study periods
  Interventions: Drug: Phenylephrine HCl Extended Release
- Phenylephrine HCl Extended Release - Fed (Experimental): Single dose phenylephrine HCl extended release tablet administered after a high-fat, high-calorie breakfast on Day 1 in one of four study periods
  Interventions: Drug: Phenylephrine HCl Extended Release
- Phenylephrine HCl Immediate Release - Fasted (Active Comparator): Three single doses of phenylephrine HCl immediate release tablet four hours apart, with the first dose administered under fasted conditions on Day 1 in one of four study periods
  Interventions: Drug: Phenylephrine HCl Immediate Release
- Phenylephrine HCl Immediate Release - Fed (Active Comparator): Three single doses of phenylephrine HCl immediate release tablet four hours apart, with the first dose administered after a high-fat, high-calorie breakfast on Day 1 in one of four study periods
  Interventions: Drug: Phenylephrine HCl Immediate Release

INTERVENTIONS:
Drug: Phenylephrine HCl Extended Release — One phenylephrine HCl 30 mg extended release tablet orally
  Arms: Phenylephrine HCl Extended Release - Fasted; Phenylephrine HCl Extended Release - Fed
Drug: Phenylephrine HCl Immediate Release — One phenylephrine HCl 10 mg immediate release tablet every 4 hours for three doses
  Arms: Phenylephrine HCl Immediate Release - Fasted; Phenylephrine HCl Immediate Release - Fed

SUMMARY:
This study will assess the food-effect bioavailability of an extended release formulation of phenylephrine HCl and its bioequivalence to the marketed immediate release phenylephrine HCl product.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* Female participants must not be pregnant
* Agrees to use two acceptable methods of birth control throughout the study
* Agrees not to take monoamine oxidase inhibitor (MAOI) for 2 weeks prior to, during, and 2 weeks after the end of the study

Exclusion Criteria:

* Any significant medical condition which is a contraindication to the use of phenylephrine HCl, might interfere with the study, or requires treatment expected to affect blood pressure
* Any infectious disease within 4 weeks prior to initial treatment administration
* History of malignancy, except basal cell carcinoma
* Cannot comply with requirement to abstain from the use of any drugs (except acetaminophen or herbal/vitamin supplements) within 14 days prior to study and alcohol or xanthine-containing substances (coffee, chocolate) within 72 hours prior to study
* Received an investigational drug within thirty days prior to study drug dosing
* Known or apparent current or former drug addicts or alcoholics
* Positive for Human Immunodeficiency Virus (HIV) antibody, hepatitis B surface antigen, or hepatitis C antibody
* Cannot accept a high-fat, high-calorie breakfast
* Known allergy or intolerance to phenylephrine HCl
* Have used phenylephrine-containing product within 2 weeks prior to study start
* Have smoked tobacco, used tobacco products, or used a nicotine-containing smoking cessation aid within the past 6 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of phenylephrine | 0 hours to time of maximum observed plasma concentration of phenylephrine (blood samples will be collected up to 24 hours after first administration of study treatment)
Time to Cmax (Tmax) of phenylephrine | 0 hours to time of maximum observed plasma concentration of phenylephrine (blood samples will be collected up to 24 hours after first administration of study treatment)
Area under the concentration versus time curve from time 0 to the last measurable concentration (AUC[0-t]) | 0 hours to time of last measurable plasma concentration of phenylephrine (blood samples will be collected up to 24 hours after first administration of study treatment)
Area under the concentration versus time curve from time 0 to infinity (AUC[0-∞]) | 0 hours to time of last measurable plasma concentration of phenylephrine (blood samples will be collected up to 24 hours after first administration of study treatment)
Terminal rate constant (λz) | 0 hours to time of last measurable plasma concentration of phenylephrine (blood samples will be collected up to 24 hours after first administration of study treatment)
Terminal elimination half-life (t1/2) | 0 hours to t1/2 of phenylephrine (blood samples will be collected up to 24 hours after first administration of study treatment)